CLINICAL TRIAL: NCT02041533
Title: An Open-Label, Randomized, Phase 3 Trial of Nivolumab Versus Investigator's Choice Chemotherapy as First-Line Therapy for Stage IV or Recurrent PD-L1+ Non-Small Cell Lung Cancer
Brief Title: An Open-Label, Randomized, Phase 3 Trial of Nivolumab Versus Investigator's Choice Chemotherapy as First-Line Therapy for Stage IV or Recurrent PD-L1+ Non-Small Cell Lung Cancer (CheckMate 026)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Collaborators: Ono Pharmaceutical Co. Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA209-026; 2012-004502-93 (EudraCT Number)
Record Dates: First submitted 2014-01-19; First posted 2014-01-22 (Estimated); Results first posted 2017-07-26 (Actual); Last update posted 2023-03-02 (Actual); Status verified 2023-02

CONDITIONS: Stage IV or Recurrent Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Nivolumab; Gemcitabine; Cisplatin; Carboplatin; Paclitaxel; Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A: Nivolumab subjects (Experimental): Nivolumab solution for Injection 3 mg/kg Intravenous every 2 weeks until disease progression, discontinuation due to unacceptable toxicity, withdrawal of consent or study closure
  Interventions: Biological: Nivolumab
- Arm B: Investigator's Choice Chemotherapy (Active Comparator): Investigator's Choice Chemotherapy administered in 3-week cycles up to a maximum of 6 cycles of Intravenous injection until disease progression, unacceptable toxicity or completion of the 6 cycles, whichever comes first
  Squamous subjects:
  * Gemcitabine 1250 mg/mg(2) administered on Day 1 and Day 8 with Cisplatin 75 mg/m(2) administered on Day 1 of each cycle; or
  * Gemcitabine 1000 mg/mg(2) administered on Day 1 and Day 8 with Carboplatin (AUC 5) administered on Day 1 of each cycle; or
  * Paclitaxel 200 mg/m(2) with Carboplatin (AUC 6) administered on Day 1 of each cycle
  Non-Squamous subjects:
  * Pemetrexed 500 mg/m(2) with Cisplatin 75 mg/m(2) administered on Day 1 of each cycle
  * Pemetrexed 500 mg/m(2) Carboplatin (AUC 6) administered on Day 1 of each cycle
  Optional crossover:
  * Nivolumab solution for Injection 3 mg/kg Intravenous every 2 weeks until disease progression, discontinuation due to toxicity, withdrawal of consent or study closure
  Interventions: Biological: Nivolumab; Drug: Gemcitabine; Drug: Cisplatin; Drug: Carboplatin; Drug: Paclitaxel; Drug: Pemetrexed

INTERVENTIONS:
Biological: Nivolumab
  Other Names: BMS-936558; MDX-1106
Drug: Gemcitabine
  Other Names: Gemzar
  Arms: Arm B: Investigator's Choice Chemotherapy
Drug: Cisplatin
  Other Names: Platinol
  Arms: Arm B: Investigator's Choice Chemotherapy
Drug: Carboplatin
  Other Names: Paraplatin
  Arms: Arm B: Investigator's Choice Chemotherapy
Drug: Paclitaxel
  Other Names: Taxol
  Arms: Arm B: Investigator's Choice Chemotherapy
Drug: Pemetrexed
  Other Names: Alimta
  Arms: Arm B: Investigator's Choice Chemotherapy

SUMMARY:
The purpose of this study is to show that Nivolumab will improve progression free survival in subjects with strongly Stage IV or Recurrent PD-L1+ non-small cell lung cancer when compared to chemotherapy

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) ≤ 1
* Histologically confirmed Stage IV, or Recurrent NSCLC with no prior systemic anticancer therapy
* Measurable disease by computed tomography (CT) or magnetic resonance imaging (MRI) per response evaluation criteria in solid tumors version (RECIST) 1.1 criteria
* PD-L1+ on immunohistochemistry testing performed by central lab
* Men and women, ages ≥ 18 years of age

Exclusion Criteria:

* Known epidermal growth factor receptor (EGFR) mutations which are sensitive to available targeted inhibitor therapy
* Known anaplastic lymphoma kinase (ALK) translocations
* Untreated central nervous system (CNS) metastases
* Previous malignancies
* Active, known or suspected autoimmune disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 541 (Actual)
Dates: Start 2014-03-27 (Actual); Primary Completion 2016-07-01 (Actual); Study Completion 2022-05-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (141):
- United States (36):
  - Southern Cancer Center, Inc., Mobile, Alabama
  - Banner MD Anderson Cancer Center, Gilbert, Arizona
  - Local Institution - 0034, Tucson, Arizona
  - Local Institution - 0016, Stanford, California
  - University Of Colorado Hosp, Aurora, Colorado
  - Local Institution - 0020, New Haven, Connecticut
  - Local Institution - 0030, Miami, Florida
  - Local Institution - 0033, Ocala, Florida
  - H. Lee Moffitt Cancer Center, Tampa, Florida
  - Local Institution - 0010, Atlanta, Georgia
  - Northwest Georgia Oncology Center, P.C., Marietta, Georgia
  - Local Institution - 0037, Chicago, Illinois
  - Local Institution - 0014, Lexington, Kentucky
  - Crescent City Research Consortium, LLC, Marrero, Louisiana
  - Local Institution - 0024, Baltimore, Maryland
  - Local Institution - 0036, Boston, Massachusetts
  - Local Institution - 0070, Boston, Massachusetts
  - Roswell Park Cancer Institute, Buffalo, New York
  - Local Institution - 0009, New York, New York
  - Local Institution - 0005, New York, New York
  - University Of North Carolina At Chapel Hill, Chapel Hill, North Carolina
  - Local Institution - 0003, Durham, North Carolina
  - Local Institution - 0012, Cleveland, Ohio
  - Local Institution - 0027, Columbus, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - Local Institution - 0007, Allentown, Pennsylvania
  - Local Institution - 0054, Philadelphia, Pennsylvania
  - Local Institution - 0002, Philadelphia, Pennsylvania
  - Local Institution - 0018, Pittsburgh, Pennsylvania
  - Local Institution - 0011, Charleston, South Carolina
  - Local Institution - 0038, Greenville, South Carolina
  - Local Institution - 0008, Nashville, Tennessee
  - Local Institution - 0006, Dallas, Texas
  - Local Institution - 0023, Houston, Texas
  - Cancer Centers of South Texas, San Antonio, Texas
  - Local Institution - 0029, Yakima, Washington
- Argentina (5):
  - Local Institution - 0051, Berazategui, Buenos Aires
  - Local Institution - 0049, Capital Federal, Buenos Aires
  - Local Institution - 0052, Ciudad Autonoma de Buenos Aire, Buenos Aires
  - Local Institution - 0048, Córdoba
  - Local Institution - 0050, Córdoba
- Australia (5):
  - Local Institution - 0090, Camperdown, New South Wales
  - Local Institution - 0091, Brisbane, Queensland
  - Local Institution - 0071, Elizabeth Vale, South Australia
  - Local Institution - 0072, Fitzroy, Victoria
  - Local Institution - 0104, Heidelberg, Victoria
- Austria (2):
  - Local Institution - 0087, Vienna
  - Local Institution - 0088, Wels
- Belgium (4):
  - Local Institution - 0044, Brussels
  - Local Institution - 0055, Edegem
  - Local Institution - 0056, Ghent
  - Local Institution - 0062, Leuven
- Brazil (3):
  - Local Institution - 0134, Ijuí, Rio Grande do Sul
  - Local Institution - 0133, Porto Alegre, Rio Grande do Sul
  - Local Institution - 0135, Barretos, São Paulo
- Canada (5):
  - Local Institution - 0086, Calgary, Alberta
  - Local Institution - 0115, Hamilton, Ontario
  - Local Institution - 0113, Toronto, Ontario
  - Local Institution - 0110, Montreal, Quebec
  - Local Institution - 0109, Rimouski, Quebec
- Czechia (4):
  - Local Institution - 0059, Olomouc
  - Local Institution - 0061, Ostrava - Poruba
  - Local Institution - 0058, Prague
  - Local Institution - 0060, Ústí nad Labem
- Finland (3):
  - Local Institution - 0120, Helsinki
  - Local Institution - 0119, Tampere
  - Local Institution - 0118, Vaasa
- France (6):
  - Local Institution - 0123, Caen
  - Local Institution - 0105, Lille
  - Local Institution - 0102, Marseille
  - Local Institution - 0167, Pontoise
  - Local Institution - 0100, Rennes
  - Local Institution - 0140, Strasbourg
- Germany (6):
  - Local Institution - 0074, Bamberg
  - Local Institution - 0063, Cologne
  - Local Institution - 0065, Großhansdorf
  - Local Institution - 0064, Heidelberg
  - Local Institution - 0066, Stuttgart
  - Local Institution - 0092, Wiesbaden
- Greece (2):
  - Local Institution - 0073, Heraklion, Crete
  - Local Institution - 0075, Athens
- Hungary (3):
  - Local Institution - 0126, Budapest
  - Local Institution - 0116, Debrecen
  - Local Institution - 0094, Mátraháza
- Italy (6):
  - Local Institution - 0084, Avellino
  - Local Institution - 0079, Livorno
  - Local Institution - 0143, Milan
  - Local Institution - 0142, Napoli
  - Local Institution - 0083, Perugia
  - Local Institution - 0082, Terni
- Japan (18):
  - Local Institution - 0146, Nagoya, Aichi-ken
  - Local Institution - 0161, Nagoya, Aichi-ken
  - Local Institution - 0148, Matsuyama, Ehime
  - Local Institution - 0153, Kobe, Hyōgo
  - Local Institution - 0144, Natori-shi, Miyagi
  - Local Institution - 0151, Niigata, Niigata
  - Local Institution - 0166, Habikino-shi, Osaka
  - Local Institution - 0147, Miyakojima-ku, Osaka
  - Local Institution - 0145, Ōsaka-sayama, Osaka
  - Local Institution - 0152, Sakai, Osaka
  - Local Institution - 0150, Kitaadachi-gun, Saitama
  - Local Institution - 0149, Sunto-gun, Shizuoka
  - Local Institution - 0154, Chuo-ku, Tokyo
  - Local Institution - 0159, Akashi, Hyogo
  - Local Institution - 0162, Ota, Gunma
  - Local Institution - 0165, Sapporo, Hokkaido
  - Local Institution - 0160, Tokyo
  - Local Institution - 0158, Wakayama
- Mexico (3):
  - Local Institution - 0122, Guadalajara, Jalisco
  - Local Institution - 0117, Mexico City, Mexico City
  - Local Institution - 0124, Mérida, Yucatán
- Netherlands (3):
  - Local Institution - 0045, Amsterdam
  - Local Institution - 0057, Groningen
  - Local Institution - 0046, Rotterdam
- Poland (5):
  - Local Institution - 0114, Bydgoszcz
  - Local Institution - 0131, Krakow
  - Local Institution - 0139, Lodz
  - Local Institution - 0089, Warsaw
  - Local Institution - 0093, Wodzisław Śląski
- Romania (3):
  - Local Institution - 0068, Cluj-Napoca
  - Local Institution - 0067, Cluj-Napoca
  - Local Institution - 0069, Ploieşti
- South Korea (3):
  - Local Institution - 0155, Gangnam-gu
  - Local Institution - 0164, Seoul
  - Local Institution - 0163, Seoul
- Spain (6):
  - Local Institution - 0040, Barcelona
  - Local Institution - 0041, Las Palmas de Gran Canaria
  - Local Institution - 0047, Madrid
  - Local Institution - 0042, Málaga
  - Local Institution - 0039, Seville
  - Local Institution - 0043, Valencia
- Sweden (2):
  - Local Institution - 0127, Stockholm
  - Local Institution - 0125, Uppsala
- Switzerland (3):
  - Local Institution - 0076, Chur
  - Local Institution - 0077, Lausanne
  - Local Institution - 0078, Zurich
- Local Institution - 0157, Taipei, Taiwan
- Local Institution - 0130, Kayseri, Turkey (Türkiye)
- United Kingdom (3):
  - Local Institution - 0098, London, Greater London
  - Local Institution - 0097, Manchester, Greater Manchester
  - Local Institution - 0053, Leeds, Yorkshire

REFERENCES:
- [Derived] Mason M, Lapuente-Santana O, Halkola AS, Wang W, Mall R, Xiao X, Kaufman J, Fu J, Pfeil J, Banerjee J, Chung V, Chang H, Chasalow SD, Lin HY, Chai R, Yu T, Finotello F, Mirtti T, Mayranpaa MI, Bao J, Verschuren EW, Ahmed EI, Ceccarelli M, Miller LD, Monaco G, Hendrickx WRL, Sherif S, Yang L, Tang M, Gu SS, Zhang W, Zhang Y, Zeng Z, Das Sahu A, Liu Y, Yang W, Bedognetti D, Tang J, Eduati F, Laajala TD, Geese WJ, Guinney J, Szustakowski JD, Vincent BG, Carbone DP. A community challenge to predict clinical outcomes after immune checkpoint blockade in non-small cell lung cancer. J Transl Med. 2024 Feb 21;22(1):190. doi: 10.1186/s12967-023-04705-3. PMID 38383458
- [Derived] Carbone DP, Reck M, Paz-Ares L, Creelan B, Horn L, Steins M, Felip E, van den Heuvel MM, Ciuleanu TE, Badin F, Ready N, Hiltermann TJN, Nair S, Juergens R, Peters S, Minenza E, Wrangle JM, Rodriguez-Abreu D, Borghaei H, Blumenschein GR Jr, Villaruz LC, Havel L, Krejci J, Corral Jaime J, Chang H, Geese WJ, Bhagavatheeswaran P, Chen AC, Socinski MA; CheckMate 026 Investigators. First-Line Nivolumab in Stage IV or Recurrent Non-Small-Cell Lung Cancer. N Engl J Med. 2017 Jun 22;376(25):2415-2426. doi: 10.1056/NEJMoa1613493. PMID 28636851
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Nivolumab: Nivolumab 3mg/kg IV infusion, every 2 weeks until disease progression or unacceptable toxicity
- Investigator Choice of Chemotherapy: Administered in 3-week cycles for up to 6 cycles:
  Squamous:
  * gemcitabine (1250 mg/mg2) with cisplatin (75 mg/m2); or
  * gemcitabine (1000 mg/m2) with carboplatin (AUC 5); or
  * paclitaxel (200 mg/m2) with carboplatin (AUC 6)
  Non-Squamous:
  * pemetrexed (500 mg/m2) with cisplatin (75 mg/m2); or
  * pemetrexed (500 mg/m2) with carboplatin (AUC 6) Subjects who discontinued cisplatin could be switched to gemcitabine/carboplatin for the remainder of the platinum doublet cycles (up to 6 cycles in total). Participants who progressed on or after chemotherapy could be eligible to receive optional crossover nivolumab 3 mg/kg administered every 2 weeks until disease progression, discontinuation due to unacceptable toxicity, withdrawal of consent or study closure.
Period: Pre-Treatment Period
Arm/Group | Nivolumab | Investigator Choice of Chemotherapy
Started (Started = Participants Randomized) | 271 | 270
Completed (Completed = Participants Treated) | 267 | 263
Not Completed | 4 | 7
Not completed — Disease Progression | 1 | 1
Not completed — Participant Withdrew Consent | 0 | 5
Not completed — Participant no Longer Meets Study Criteria | 3 | 1
Period: Treatment Period
Arm/Group | Nivolumab | Investigator Choice of Chemotherapy
Started | 267 | 263
Received Optional Nivolumab (Participants in the Investigator Choice Arm who progressed on or after chemotherapy could be eligible to receive optional crossover nivolumab.) | 0 | 159
Completed | 0 | 28
Not Completed | 267 | 235
Not completed — Disease progression | 189 | 146
Not completed — Study drug toxicity | 30 | 34
Not completed — Death | 1 | 0
Not completed — Adverse event unrelated to study drug | 22 | 23
Not completed — Participant request to discontinue study treatment | 12 | 9
Not completed — Participant withdrew consent | 2 | 2
Not completed — Maximum clinical benefit | 0 | 18
Not completed — Poor/Non-compliance | 1 | 0
Not completed — Administrative reason by sponsor | 1 | 0
Not completed — Other reasons | 9 | 2
Not completed — Not Reported | 0 | 1

BASELINE CHARACTERISTICS:
Population: All randomized participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Nivolumab | Investigator Choice of Chemotherapy | Total
Number analyzed (Participants) | 271 | 270 | 541
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.8 (10.25) | 63.4 (9.63) | 63.1 (9.94)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 87 | 122 | 209
  Male | 184 | 148 | 332
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 3 | 7
  Not Hispanic or Latino | 141 | 139 | 280
  Unknown or Not Reported | 126 | 128 | 254
Race/Ethnicity, Customized [Number; unit: Participants] — Race
  Participants
    White | 228 | 242 | 470
    Black or African American | 6 | 10 | 16
    Asian | 30 | 17 | 47
    American Indian or Alaska Native | 1 | 0 | 1
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Other | 6 | 1 | 7

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival in Participants With PD-L1 Expression >= 5%
Description: Progression-Free Survival (PFS) was defined as the time between the date of randomization and the first date of documented tumor progression, as determined by the Independent Radiology Review Committee (IRRC) per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1, or death due to any cause, whichever occurs first. Participants who die without a reported progression were considered to have progressed on the date of their death. Participants who did not progress or die were censored on the date of their last evaluable tumor assessment. Participants who did not have any on-study tumor assessments and did not die were censored on the day they were randomized. Participants who received subsequent anti-cancer therapy prior to documented progression were censored at the last evaluable tumor assessment prior to the initiation of new therapy.
Time Frame: From date of randomization until date of documented tumor progression (assessed up to August 2016, approximately 28 months)
Population: All randomized participants with PD-L1 expression levels >= 5%
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Nivolumab | Investigator Choice of Chemotherapy
Number analyzed (Participants) | 211 | 212
Months | 4.21 [2.96 to 5.55] | 5.88 [5.42 to 6.93]
Statistical Analysis 1: Comparison: Nivolumab vs Investigator Choice of Chemotherapy; Test type: Superiority or Other; p = 0.2511, Log Rank; Log-rank test stratified by histology (squamous vs. non-squamous) as entered into the IVRS; Hazard Ratio (HR) = 1.15, 95% CI 2-sided [0.91 to 1.45] — Stratified Cox proportional hazard model. Hazard ratio of nivolumab to investigator's choice chemotherapy

2. Secondary Outcome: Progression-Free Survival in All Randomized Participants
Description: as for outcome 1
Time Frame: as for outcome 1
Population: All randomized participants
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Nivolumab | Investigator Choice of Chemotherapy
Number analyzed (Participants) | 271 | 270
Months | 4.21 [3.06 to 5.52] | 5.82 [5.42 to 6.90]
Statistical Analysis 1: Comparison: Nivolumab vs Investigator Choice of Chemotherapy; Test type: Superiority or Other; Hazard Ratio (HR) = 1.17, 95% CI 2-sided [0.95 to 1.43] — Stratified Cox proportional hazard model. Hazard ratio of nivolumab to investigator's choice chemotherapy

3. Secondary Outcome: Overall Survival in Participants With PD-L1 Expression >= 5%
Description: Overall Survival (OS) was defined as the time from randomization to the date of death. A participant who had not died was censored at the last known alive date. OS was censored at the date of randomization for participants who were randomized but had no follow-up.
Time Frame: From date of randomization to date of death (up to approximately 89 months)
Population: All randomized participants with PD-L1 expression >= 5%
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Nivolumab | Investigator Choice of Chemotherapy
Number analyzed (Participants) | 211 | 212
Months | 14.36 [11.66 to 17.08] | 13.21 [10.81 to 17.28]
Statistical Analysis 1: Comparison: Nivolumab vs Investigator Choice of Chemotherapy; Test type: Superiority; Hazard Ratio (HR) = 0.97, 95% CI 2-sided [0.79 to 1.20] — Stratified Cox proportional hazard model. Hazard ratio of nivolumab to investigator's choice chemotherapy

4. Secondary Outcome: Overall Survival in All Randomized Participants
Description: as for outcome 3
Time Frame: From date of randomization to date of death (up to approximately 89 months)
Population: All randomized participants
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Nivolumab | Investigator Choice of Chemotherapy
Number analyzed (Participants) | 271 | 270
Months | 13.73 [11.76 to 15.41] | 13.80 [11.01 to 16.99]
Statistical Analysis 1: Comparison: Nivolumab vs Investigator Choice of Chemotherapy; Test type: Superiority; Hazard Ratio (HR) = 1.03, 95% CI 2-sided [0.86 to 1.24] — Stratified Cox proportional hazard model. Hazard ratio of nivolumab to investigator's choice chemotherapy

5. Secondary Outcome: Objective Response Rate (ORR) in Participants With PD-L1 Expression >= 5%
Description: ORR was defined as the proportion of randomized participants who achieved a Best Overall Response (BOR) of CR or PR using the RECIST v1.1 criteria per Independent Radiology Review Committee (IRRC) assessment. BOR was defined as the best response designation recorded between the date of randomization and the date of objectively documented progression or start of subsequent anti-cancer therapy, whichever occurred first. For participants without documented progression or subsequent therapy, all available response designations contributed to the BOR assessment. For participants who continued treatment beyond progression, BOR was determined from response designations recorded up to the time of initial progression. CR= Disappearance of all evidence of disease, confirmed by PET scan; PR= Regression of measureable disease and no new sites; Stable Disease (SD)= Failure to attain CR/PR or PD; Progressive Disease (PD)= Any new lesion or increase by >=50% of previously involved sites from nadir.
Time Frame: From date of randomization until date of documented tumor progression or subsequent anti-cancer therapy, whichever occurs first (assessed up to August 2016, approximately 28 months)
Population: All randomized participants with PD-L1 expression >= 5%
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Nivolumab | Investigator Choice of Chemotherapy
Number analyzed (Participants) | 211 | 212
Percentage of participants | 26.1 [20.3 to 32.5] | 33.5 [27.2 to 40.3]
Statistical Analysis 1: Comparison: Nivolumab vs Investigator Choice of Chemotherapy; Test type: Superiority or Other; Odds Ratio (OR) = 0.70, 95% CI 2-sided [0.46 to 1.06] — Stratified by histology (squamous vs.non-squamous) at randomization. Strata adjusted odds ratio (Nivolumab over investigator choice of chemotherapy) using Mantel-Haenszel method

6. Secondary Outcome: Disease-related Symptom Improvement Rate by Week 12
Description: The Lung Cancer Symptom Score (LCSS) is a validated instrument designed to assess the impact of treatment on disease-related symptoms. It consists of 6 symptom-specific questions related to dyspnea, cough, fatigue, pain, hemoptysis and anorexia plus 3 summary items: symptom distress, interference with activity, and global HRQoL. The degree of impairment was recorded on a 100 mm visual analogue scale with scores from 0 to 100 with zero representing the best score. Disease-related symptom improvement rate by Week 12 is defined as the proportion of all randomized (all PD-L1+) participants who had 10 points or more decrease from baseline in average symptom burden index score at any time between randomization and Week 12.
Time Frame: From date of randomization to week 12
Population: All randomized participants
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Nivolumab | Investigator Choice of Chemotherapy
Number analyzed (Participants) | 271 | 270
Percentage of participants | 35.4 [29.7 to 41.4] | 33.7 [28.1 to 39.7]

ADVERSE EVENTS:
Time Frame: Participants were assessed for All-Cause Mortality from the date of their randomization until study completion (up to approximately 89 months). SAEs and Other AEs were assessed from their first dose to 100 days following their last dose (up to approximately 89 months).
Description: The number at Risk for All-Cause Mortality represents all Randomized Participants. The number at risk for Serious Adverse Events and Other (Not Including Serious) Adverse Events represents all participants that received at least 1 dose of study medication.
Groups:
- Post Chemotherapy Optional Nivolumab: Participants from the Investigator Choice Arm who progressed during Post-Chemotherapy Phase could receive crossover nivolumab treatment after disease progression. These participants received Nivolumab 3 mg/kg IV infusion every 2 weeks until disease progression, discontinuation due to unacceptable toxicity, withdrawal of consent or study closure.
Arm/Group | Nivolumab | Investigator Choice of Chemotherapy | Post Chemotherapy Optional Nivolumab
All-Cause Mortality (participants affected / at risk) | 233/271 | 92/270 | 136/159
Serious Adverse Events (participants affected / at risk) | 195/267 | 203/263 | 110/159
Other Adverse Events (participants affected / at risk) | 245/267 | 252/263 | 137/159
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nivolumab (N=267) | Investigator Choice of Chemotherapy (N=263) | Post Chemotherapy Optional Nivolumab (N=159)
Anaemia (Blood and lymphatic system disorders) | 1 | 16 | 2
Anaemia of malignant disease (Blood and lymphatic system disorders) | 0 | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 3 | 7 | 1
Haemolytic anaemia (Blood and lymphatic system disorders) | 2 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 4 | 1
Pancytopenia (Blood and lymphatic system disorders) | 1 | 3 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 6 | 0
Acute coronary syndrome (Cardiac disorders) | 3 | 1 | 0
Acute left ventricular failure (Cardiac disorders) | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 6 | 3
Atrial flutter (Cardiac disorders) | 0 | 3 | 2
Atrial tachycardia (Cardiac disorders) | 0 | 1 | 0
Bradycardia (Cardiac disorders) | 0 | 1 | 1
Cardiac arrest (Cardiac disorders) | 1 | 0 | 0
Cardiac failure (Cardiac disorders) | 2 | 4 | 3
Cardiac failure acute (Cardiac disorders) | 1 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 2 | 1 | 0
Cardiac tamponade (Cardiac disorders) | 1 | 0 | 0
Cardiovascular disorder (Cardiac disorders) | 0 | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 7 | 4
Myocardial ischaemia (Cardiac disorders) | 1 | 1 | 0
Pericardial effusion (Cardiac disorders) | 0 | 2 | 1
Pericarditis constrictive (Cardiac disorders) | 0 | 1 | 0
Sinus bradycardia (Cardiac disorders) | 1 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 1 | 0
Tornwaldt cyst (Congenital, familial and genetic disorders) | 1 | 0 | 0
Adrenal insufficiency (Endocrine disorders) | 4 | 4 | 2
Hypothyroidism (Endocrine disorders) | 0 | 2 | 2
Angle closure glaucoma (Eye disorders) | 0 | 1 | 0
Cataract (Eye disorders) | 1 | 0 | 0
Exophthalmos (Eye disorders) | 0 | 1 | 0
Glaucoma (Eye disorders) | 0 | 1 | 0
Ophthalmic vein thrombosis (Eye disorders) | 0 | 1 | 1
Optic nerve disorder (Eye disorders) | 0 | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 4 | 1
Ascites (Gastrointestinal disorders) | 1 | 0 | 0
Colitis (Gastrointestinal disorders) | 4 | 3 | 3
Constipation (Gastrointestinal disorders) | 2 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 7 | 6 | 4
Dysphagia (Gastrointestinal disorders) | 1 | 1 | 0
Enteritis (Gastrointestinal disorders) | 0 | 1 | 1
Gastritis (Gastrointestinal disorders) | 0 | 1 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 2 | 1
Ileus (Gastrointestinal disorders) | 0 | 3 | 0
Large intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0
Large intestine perforation (Gastrointestinal disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 4 | 5 | 1
Oesophagitis (Gastrointestinal disorders) | 1 | 0 | 0
Small intestinal haemorrhage (Gastrointestinal disorders) | 0 | 2 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 2 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 1 | 1
Vomiting (Gastrointestinal disorders) | 4 | 5 | 1
Asthenia (General disorders) | 2 | 0 | 0
Catheter site pain (General disorders) | 0 | 1 | 0
Chest pain (General disorders) | 2 | 2 | 0
Death (General disorders) | 1 | 0 | 0
Fatigue (General disorders) | 2 | 8 | 3
General physical health deterioration (General disorders) | 4 | 6 | 4
Illness (General disorders) | 1 | 0 | 0
Localised oedema (General disorders) | 0 | 1 | 1
Multiple organ dysfunction syndrome (General disorders) | 2 | 0 | 0
Oedema peripheral (General disorders) | 1 | 0 | 0
Pain (General disorders) | 1 | 3 | 1
Performance status decreased (General disorders) | 0 | 2 | 0
Pyrexia (General disorders) | 7 | 9 | 6
Sudden death (General disorders) | 1 | 0 | 0
Bile duct stenosis (Hepatobiliary disorders) | 0 | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1 | 1
Cholecystitis acute (Hepatobiliary disorders) | 2 | 1 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 1
Cholestasis (Hepatobiliary disorders) | 1 | 1 | 0
Drug-induced liver injury (Hepatobiliary disorders) | 0 | 1 | 1
Gallbladder obstruction (Hepatobiliary disorders) | 0 | 1 | 0
Hepatic failure (Hepatobiliary disorders) | 1 | 1 | 0
Hepatitis (Hepatobiliary disorders) | 1 | 1 | 1
Hepatitis acute (Hepatobiliary disorders) | 1 | 0 | 0
Hypertransaminasaemia (Hepatobiliary disorders) | 1 | 0 | 0
Jaundice (Hepatobiliary disorders) | 0 | 1 | 0
Hypersensitivity (Immune system disorders) | 3 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 2 | 1
Appendicitis perforated (Infections and infestations) | 0 | 1 | 0
Bronchitis (Infections and infestations) | 2 | 3 | 1
Cellulitis (Infections and infestations) | 0 | 1 | 0
Diverticulitis (Infections and infestations) | 1 | 0 | 0
Erysipelas (Infections and infestations) | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 1 | 1
Herpes virus infection (Infections and infestations) | 0 | 1 | 0
Infection (Infections and infestations) | 0 | 1 | 1
Influenza (Infections and infestations) | 0 | 1 | 0
Localised infection (Infections and infestations) | 0 | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 2 | 1 | 1
Nasopharyngitis (Infections and infestations) | 1 | 0 | 0
Norovirus infection (Infections and infestations) | 1 | 0 | 0
Oral candidiasis (Infections and infestations) | 0 | 1 | 1
Peritonitis (Infections and infestations) | 0 | 1 | 0
Pleural infection (Infections and infestations) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 21 | 26 | 8
Pneumonia aspiration (Infections and infestations) | 1 | 0 | 0
Pneumonia bacterial (Infections and infestations) | 1 | 1 | 0
Post procedural infection (Infections and infestations) | 0 | 1 | 1
Pulmonary sepsis (Infections and infestations) | 0 | 1 | 0
Respiratory tract infection (Infections and infestations) | 1 | 2 | 1
Sepsis (Infections and infestations) | 5 | 5 | 3
Septic shock (Infections and infestations) | 1 | 1 | 0
Skin infection (Infections and infestations) | 0 | 2 | 0
Subcutaneous abscess (Infections and infestations) | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 3 | 2 | 2
Vascular device infection (Infections and infestations) | 0 | 1 | 1
Wound infection (Infections and infestations) | 0 | 1 | 0
Compression fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 1 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 2 | 0
Hip fracture (Injury, poisoning and procedural complications) | 2 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 2 | 0 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 1 | 1
Kyphosis postoperative (Injury, poisoning and procedural complications) | 0 | 1 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Procedural pneumothorax (Injury, poisoning and procedural complications) | 1 | 0 | 0
Radiation necrosis (Injury, poisoning and procedural complications) | 1 | 0 | 0
Radiation pneumonitis (Injury, poisoning and procedural complications) | 1 | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 1 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Vascular procedure complication (Injury, poisoning and procedural complications) | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 5 | 1 | 1
Aspartate aminotransferase increased (Investigations) | 6 | 2 | 2
Blood alkaline phosphatase increased (Investigations) | 1 | 0 | 0
Blood bilirubin increased (Investigations) | 1 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 1 | 1
Blood creatinine increased (Investigations) | 2 | 1 | 0
C-reactive protein increased (Investigations) | 0 | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 2 | 0 | 0
General physical condition abnormal (Investigations) | 1 | 0 | 0
Haemoglobin decreased (Investigations) | 0 | 1 | 0
Transaminases increased (Investigations) | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 4 | 5 | 3
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 3 | 3 | 3
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 2 | 2
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 1 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 5 | 4 | 2
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 3 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Osteolysis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1
Pathological fracture (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Polyarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8 | 2 | 1
Chronic myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Follicular lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Haemangioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Intestinal metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 2
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 69 | 95 | 55
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 5 | 3
Mesothelioma malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 8 | 6
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Metastases to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0 | 0
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2 | 0
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1 | 1
Non-small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Pericardial effusion malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 2 | 0
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 2 | 1
Aphasia (Nervous system disorders) | 1 | 0 | 0
Ataxia (Nervous system disorders) | 0 | 2 | 1
Cerebral infarction (Nervous system disorders) | 0 | 1 | 1
Cerebrovascular accident (Nervous system disorders) | 2 | 1 | 0
Cubital tunnel syndrome (Nervous system disorders) | 0 | 1 | 1
Depressed level of consciousness (Nervous system disorders) | 1 | 0 | 0
Epilepsy (Nervous system disorders) | 1 | 0 | 0
Headache (Nervous system disorders) | 2 | 0 | 0
IIIrd nerve paresis (Nervous system disorders) | 0 | 1 | 1
Ischaemic stroke (Nervous system disorders) | 1 | 1 | 0
Loss of consciousness (Nervous system disorders) | 0 | 1 | 0
Malignant spinal cord compression (Nervous system disorders) | 1 | 0 | 0
Muscle spasticity (Nervous system disorders) | 1 | 0 | 0
Nervous system disorder (Nervous system disorders) | 0 | 1 | 1
Peripheral motor neuropathy (Nervous system disorders) | 0 | 1 | 1
Presyncope (Nervous system disorders) | 1 | 1 | 0
Seizure (Nervous system disorders) | 4 | 3 | 1
Spinal cord compression (Nervous system disorders) | 1 | 1 | 0
Syncope (Nervous system disorders) | 4 | 3 | 0
VIth nerve paresis (Nervous system disorders) | 0 | 1 | 1
Vocal cord paralysis (Nervous system disorders) | 0 | 1 | 0
Device occlusion (Product Issues) | 0 | 1 | 1
Alcohol withdrawal syndrome (Psychiatric disorders) | 1 | 0 | 0
Confusional state (Psychiatric disorders) | 3 | 2 | 1
Disorientation (Psychiatric disorders) | 0 | 1 | 1
Mental status changes (Psychiatric disorders) | 1 | 0 | 0
Organic brain syndrome (Psychiatric disorders) | 1 | 0 | 0
Psychotic disorder (Psychiatric disorders) | 1 | 0 | 0
Suicide attempt (Psychiatric disorders) | 1 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 2 | 0 | 0
Haematuria (Renal and urinary disorders) | 1 | 1 | 1
Hydronephrosis (Renal and urinary disorders) | 0 | 1 | 1
Oliguria (Renal and urinary disorders) | 1 | 0 | 0
Renal failure (Renal and urinary disorders) | 2 | 1 | 1
Renal infarct (Renal and urinary disorders) | 0 | 1 | 0
Tubulointerstitial nephritis (Renal and urinary disorders) | 1 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 3 | 7 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 | 9 | 5
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Eosinophilic pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1
Laryngeal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Mediastinal disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 8 | 5 | 3
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 9 | 2 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 4 | 2 | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 8 | 11 | 5
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary microemboli (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 4 | 2 | 2
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Air embolism (Vascular disorders) | 1 | 0 | 0
Aortic aneurysm rupture (Vascular disorders) | 1 | 0 | 0
Circulatory collapse (Vascular disorders) | 0 | 3 | 1
Deep vein thrombosis (Vascular disorders) | 3 | 1 | 1
Embolism (Vascular disorders) | 0 | 4 | 1
Extremity necrosis (Vascular disorders) | 1 | 0 | 0
Hypotension (Vascular disorders) | 1 | 1 | 0
Iliac artery occlusion (Vascular disorders) | 0 | 1 | 0
Jugular vein thrombosis (Vascular disorders) | 1 | 0 | 0
Leriche syndrome (Vascular disorders) | 0 | 1 | 0
Lymphoedema (Vascular disorders) | 0 | 1 | 1
Peripheral artery thrombosis (Vascular disorders) | 0 | 1 | 0
Peripheral ischaemia (Vascular disorders) | 1 | 0 | 0
Superior vena cava syndrome (Vascular disorders) | 0 | 2 | 0
Vascular occlusion (Vascular disorders) | 0 | 1 | 0
Vein disorder (Vascular disorders) | 1 | 0 | 0
Venous thrombosis (Vascular disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Nivolumab (N=267) | Investigator Choice of Chemotherapy (N=263) | Post Chemotherapy Optional Nivolumab (N=159)
Anaemia (Blood and lymphatic system disorders) | 54 | 142 | 38
Leukopenia (Blood and lymphatic system disorders) | 1 | 17 | 1
Neutropenia (Blood and lymphatic system disorders) | 5 | 54 | 4
Thrombocytopenia (Blood and lymphatic system disorders) | 5 | 40 | 4
Hypothyroidism (Endocrine disorders) | 23 | 23 | 14
Lacrimation increased (Eye disorders) | 3 | 21 | 1
Abdominal pain (Gastrointestinal disorders) | 35 | 32 | 12
Abdominal pain upper (Gastrointestinal disorders) | 11 | 23 | 9
Constipation (Gastrointestinal disorders) | 65 | 84 | 24
Diarrhoea (Gastrointestinal disorders) | 84 | 82 | 29
Dry mouth (Gastrointestinal disorders) | 13 | 12 | 8
Dyspepsia (Gastrointestinal disorders) | 19 | 13 | 2
Nausea (Gastrointestinal disorders) | 86 | 149 | 36
Stomatitis (Gastrointestinal disorders) | 13 | 20 | 5
Vomiting (Gastrointestinal disorders) | 59 | 77 | 16
Asthenia (General disorders) | 26 | 41 | 13
Chest pain (General disorders) | 9 | 25 | 9
Chills (General disorders) | 18 | 18 | 6
Fatigue (General disorders) | 108 | 134 | 47
Malaise (General disorders) | 15 | 14 | 5
Mucosal inflammation (General disorders) | 7 | 23 | 3
Non-cardiac chest pain (General disorders) | 25 | 21 | 11
Oedema peripheral (General disorders) | 35 | 67 | 21
Pain (General disorders) | 14 | 12 | 9
Pyrexia (General disorders) | 37 | 55 | 22
Bronchitis (Infections and infestations) | 13 | 19 | 10
Nasopharyngitis (Infections and infestations) | 19 | 20 | 10
Pneumonia (Infections and infestations) | 25 | 23 | 9
Upper respiratory tract infection (Infections and infestations) | 24 | 24 | 9
Urinary tract infection (Infections and infestations) | 14 | 13 | 4
Fall (Injury, poisoning and procedural complications) | 15 | 11 | 5
Alanine aminotransferase increased (Investigations) | 31 | 30 | 13
Aspartate aminotransferase increased (Investigations) | 39 | 28 | 10
Blood alkaline phosphatase increased (Investigations) | 22 | 18 | 7
Blood creatinine increased (Investigations) | 13 | 34 | 17
Gamma-glutamyltransferase increased (Investigations) | 10 | 14 | 4
Lymphocyte count decreased (Investigations) | 18 | 18 | 5
Neutrophil count decreased (Investigations) | 9 | 43 | 4
Platelet count decreased (Investigations) | 12 | 38 | 1
Weight decreased (Investigations) | 42 | 37 | 12
White blood cell count decreased (Investigations) | 7 | 33 | 6
Decreased appetite (Metabolism and nutrition disorders) | 91 | 102 | 37
Dehydration (Metabolism and nutrition disorders) | 10 | 19 | 7
Hyperglycaemia (Metabolism and nutrition disorders) | 19 | 18 | 10
Hyperkalaemia (Metabolism and nutrition disorders) | 15 | 19 | 11
Hypoalbuminaemia (Metabolism and nutrition disorders) | 28 | 27 | 11
Hypokalaemia (Metabolism and nutrition disorders) | 24 | 31 | 13
Hypomagnesaemia (Metabolism and nutrition disorders) | 16 | 49 | 19
Hyponatraemia (Metabolism and nutrition disorders) | 28 | 37 | 13
Hypophosphataemia (Metabolism and nutrition disorders) | 6 | 17 | 6
Arthralgia (Musculoskeletal and connective tissue disorders) | 53 | 47 | 29
Back pain (Musculoskeletal and connective tissue disorders) | 42 | 62 | 23
Muscle spasms (Musculoskeletal and connective tissue disorders) | 9 | 14 | 10
Muscular weakness (Musculoskeletal and connective tissue disorders) | 17 | 26 | 9
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 18 | 13 | 5
Myalgia (Musculoskeletal and connective tissue disorders) | 28 | 28 | 10
Pain in extremity (Musculoskeletal and connective tissue disorders) | 23 | 31 | 11
Dizziness (Nervous system disorders) | 30 | 41 | 21
Dysgeusia (Nervous system disorders) | 14 | 25 | 7
Headache (Nervous system disorders) | 30 | 50 | 19
Neuropathy peripheral (Nervous system disorders) | 5 | 15 | 8
Peripheral sensory neuropathy (Nervous system disorders) | 7 | 24 | 7
Anxiety (Psychiatric disorders) | 17 | 18 | 12
Depression (Psychiatric disorders) | 14 | 13 | 4
Insomnia (Psychiatric disorders) | 24 | 40 | 18
Cough (Respiratory, thoracic and mediastinal disorders) | 77 | 79 | 37
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 12 | 21 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 69 | 75 | 38
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 8 | 22 | 4
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 17 | 20 | 8
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 8 | 15 | 5
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 8 | 16 | 9
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 12 | 17 | 15
Productive cough (Respiratory, thoracic and mediastinal disorders) | 30 | 25 | 8
Alopecia (Skin and subcutaneous tissue disorders) | 9 | 26 | 3
Dry skin (Skin and subcutaneous tissue disorders) | 22 | 26 | 14
Pruritus (Skin and subcutaneous tissue disorders) | 39 | 31 | 17
Rash (Skin and subcutaneous tissue disorders) | 39 | 37 | 20
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 18 | 12 | 6
Hypertension (Vascular disorders) | 18 | 19 | 8
Hypotension (Vascular disorders) | 9 | 14 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.